CLINICAL TRIAL: NCT02490358
Title: A Sputum Sample Collection Protocol for Biomarker Assay Validation in Healthy Smokers and COPD Smokers and Ex-Smokers
Brief Title: Biomarker Assay Validation in Healthy Smokers and COPD Smokers and Ex-smokers
Status: Completed | Type: Observational
Sponsor: Respivert Ltd (Industry)
Collaborators: Babraham Institute Enterprise Limited (Other)
Responsible Party: Sponsor
Other Study IDs: ENA003
Record Dates: First submitted 2015-05-26; First posted 2015-07-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Healthy smoking subjects
- 2: COPD smoking subjects
- 3: COPD ex-smoker subjects

SUMMARY:
This study will collect sputum samples from healthy smokers, COPD smokers and COPD ex-smokers to analyse biomarkers of inflammation

ELIGIBILITY:
Inclusion Criteria for Healthy Smoking Subjects

1. Must have signed an informed consent indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
2. Be between 18 and 75 years of age, inclusive, at informed consent.
3. Healthy as determined by a physician, based on medical history and physical examination.
4. Must have smoked regularly in the 12-month period preceding the screening visit and have a pack history of ≥ 5 pack years (number of pack years = number of cigarettes per day/20 x number of years smoked).

Inclusion Criteria for All COPD Subjects

1. Must have signed an informed consent indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
2. Aged between 40 and 75 years of age inclusive, at the time of signing the informed consent.
3. COPD diagnosis: Subjects with a diagnosis of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines (Celli, 2004). Symptoms must be compatible with COPD for at least 1 year prior to screening and post-bronchodilator spirometry readings at screening:

   * Post-bronchodilator FEV1/FVC ratio of <0.7
   * Post-bronchodilator FEV ≥40 % and ≤80 % of predicted normal values calculated using NHANES reference equations.

Additional Inclusion for Smoking COPD Subjects 1. Must have smoked regularly in the 12-month period preceding the screening visit and have a pack history of ≥ 5 pack years (number of pack years = number of cigarettes per day/20 x number of years smoked).

Exclusion Criteria for Healthy Smoking Subjects Any potential subject who meets any of the following criteria will be excluded from the participating study.

1. Upper or lower respiratory tract infection within 4 weeks of the screening visit.
2. Positive test for alcohol at screening.
3. Taking prescription medication in the 14 days before screening.
4. Subjects whose primary consumption of tobacco is via methods other than cigarettes (manufactured or self-rolled). Primary methods of tobacco consumption that are excluded include, but are not limited to pipes, cigars and e-cigarettes.
5. Subjects who are unable to produce a total weight of at least 0.1 grams (g) of selected sputum at screening
6. Urinary cotinine levels at screening < 30 ng/ml.
7. Subject is mentally or legally incapacitated.
8. Subject is an employee of the Sponsor or contract research organization (CRO), or a relative of an employee of the Sponsor or CRO.
9. Any other reason that the Investigator considers makes the subject unsuitable to participate.

Exclusion Criteria for COPD Subjects Any potential subject who meets any of the following criteria will be excluded from the participating study

1. Upper or lower respiratory tract infection within 4 weeks of the screening visit.
2. Positive test for alcohol at screening.
3. Subjects who are unable to produce a total weight of at least 0.1g of selected sputum at screening.
4. Subject is mentally or legally incapacitated.
5. Subject is an employee of the Sponsor or contract research organization (CRO), or a relative of an employee of the Sponsor or CRO.
6. Any other reason that the Investigator considers makes the subject unsuitable to participate.
7. A history of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
8. Taking theophylline in the 28 days before screening
9. Change in COPD medication in the 28 days before screening
10. Taking oral steroids in the 28 days before screening

Additional Exclusion Criterion for Smoking COPD Subjects

1. Subjects whose primary consumption of tobacco is via methods other than cigarettes (manufactured or self-rolled). Primary methods of tobacco consumption that are excluded include, but are not limited to pipes, cigars and e-cigarettes.
2. Urinary cotinine levels at screening < 30 ng/ml.

Additional Exclusion Criterion for Ex-Smoking COPD Subjects

1. The subject is a smoker (regular or irregular), or has smoked or used nicotine-containing products within the 6 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 20 of each of the following populations will be recruited in this study:
  * Healthy smoking subjects
  * Smoking subjects with COPD
  * Ex-smoking subjects with COPD
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Lipid metabolites in sputum cell homogenate from healthy smokers and smokers and ex-smokers with COPD. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ginny Norris, Dr, Study Director — Respivert Ltd
Locations (1):
- London, United Kingdom